CLINICAL TRIAL: NCT05389293
Title: An Open-Label, Multicenter, Single-Arm, Sequential Phase-2 Study of Mosunetuzumab Alone or With Zanubrutinib for the Treatment of Patients With Newly Diagnosed Follicular Lymphoma in Need of Systemic Therapy
Brief Title: A Study of Mosunetuzumab Alone or With Zanubrutinib in People With Follicular Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-100
Record Dates: First submitted 2022-05-23; First posted 2022-05-25 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Follicular Lymphoma; Lymphoma
Keywords: Mosunetuzumab; Follicular Lymphoma; Lymphoma; Memorial Sloan Kettering Cancer Center; 22-100
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma | interventions — zanubrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Agent Mosunetuzumab (Experimental): Participants with newly diagnosed FL in need of systemic therapy
  Interventions: Drug: Mosunetuzumab
- Mosunetuzumab + Zanubrutinib (Experimental): Participants with newly diagnosed FL in need of systemic therapy
  Interventions: Drug: Mosunetuzumab; Drug: Zanubrutinib

INTERVENTIONS:
Drug: Mosunetuzumab — During Cycle 1, Mosunetuzumab will be administered SC in a step-up dosing schedule at the dose of 5 mg on Day 1, 45 mg on Day 8, and 45 mg on Day 15). Beginning with Cycle 2, Mosunetuzumab will be administered SC at the dose of 45 mg on Day 1. Each Cycle lasts 3 weeks. After the first 8 cycles (approximately 6 months) of therapy, subjects who achieved CR will discontinue therapy, those who attained a PR will receive up to 17 doses (approximately 12 months). Subjects who achieve stable disease (SD) or who experience progressive disease (PD) will be taken off study and subsequent management will be left at the discretion of the investigator.
Drug: Zanubrutinib — In Cohort 2, Zanubrutinib is concurrently administered continuously starting on Cycle 1, Day -7 and is given for 12 months in both patients with CR and those with PR. Cohort 2 patients with evidence of circulating lymphoma cells at baseline will initiate Zanubrutinib dosing on Cycle 2 Day 1 and continue dosing for 12 months.
  Arms: Mosunetuzumab + Zanubrutinib

SUMMARY:
The purpose of this study is to find out if mosunetuzumab is an effective treatment in people with follicular lymphoma that was recently diagnosed and have not yet received any treatments for their disease.

DETAILED DESCRIPTION:
After completing enrollment of the initial 53 subjects, the researchers plan to expand the study by an additional 23 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form(s)
* Ability to comply with all the study-related procedures, in the investigator's judgement
* Age 18 years or older
* ECOG performance Status of 0, 1, or 2 [Appendix 2]
* Untreated histologically documented FL of grade 1, 2, or 3A
* Stage II bulky (noncontiguous), III, or IV bulky or high burden disease [Appendix 3]
* Need of systemic therapy as evidenced by at least one of the following criteria [also see Appendix 4]:

  * Bulky disease defined as:
  * Nodal or extranodal mass > 7cm in maximum diameter
  * ≥ 3 nodal or extranodal sites each with a diameter ≥ 3 cm
  * Presence of any of the following constitutional symptoms:
  * Fever (>38C) of unclear etiology
  * Night sweats
  * Weight loss >10% within the prior 6 months
  * Symptomatic splenomegaly
  * Mass-related symptoms
  * End-organ damage (e.g., elevated creatinine or elevated liver enzymes) that is clearly related to lymphomatous infiltration in the opinion of the investigator
  * Any one of the following cytopenias due to lymphoma:
  * Hemoglobin < 10g/dL
  * Platelets <100 x 10^9/L
  * Absolute neutrophil count (ANC) < 1.5 x 10^9/L
  * Pleural or peritoneal serous effusion (irrespective of cell content)
  * Patients with absolute lymphocytosis ≥5,000 cells/µL in the peripheral blood may be allowed to participate after discussion with the study PI
* Must be considered as a potential candidate for chemoimmunotherapy in the judgement of the treating physician
* Must have at least one bi-dimensionally measurable lesion (>1.5 cm in its largest dimension for nodal lesions, or >1.0 cm in its largest dimension for extranodal lesions by computerized tomography [CT] scan or MRI)
* Agreement to provide tumor samples as follows:

  * Agreement to undergo biopsy of a safely accessible tumor site per investigator determination prior to the first dose of mosunetuzumab.
  * Agreement to undergo repeat biopsy of the same tumor site, if safely accessible, or a different safely accessible tumor site, per investigator determination, 14 to 21 days after the first dose of mosunetuzumab.
  * Patients who are unable or unwilling to undergo either biopsy procedure may be allowed to participate in, or continue with, the study without any penalization after confirmation from the PI. Inability to undergo a new pre-treatment or an on-treatment biopsy are not considered protocol violations.
* Adequate hepatic function as follows: aspartate transaminase (AST) and alanine transaminase (ALT) levels ≤3 x upper limit of normal (ULN); total bilirubin level ≤1.5 x ULN (except with documented history of Gilbert syndrome)
* Adequate bone marrow function as follows:

  * Platelet count ≥75 x 10^9/L without transfusion within 14 days prior to first dose of mosunetuzumab;
  * ANC ≥1 x 10^9/L
  * Hemoglobin level ≥9 g/dL without transfusion within 14 days prior to the first dose of mosunetuzumab
  * Patients who do not meet criteria for bone marrow function due to marrow involvement of lymphoma and/or other disease-related cytopenias (e.g., immune thrombocytopenia) may be enrolled into the study after discussion with, and confirmation by the PI.
* Serum creatinine ≤ULN or estimated creatinine clearance ≥ 45 mL/min by Cockcroft-Gault method [see Appendix 5] or other institutional standard methods (e.g., based on nuclear medicine renal scan)
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of ≤1% per year, and agreement to refrain from donating eggs, during the treatment period and for at least 3 months after the last dose of mosunetuzumab, and 3 months after the last dose of tocilizumab (if applicable), whichever is longer.

  * A woman is considered to be of childbearing potential if she is post-menarcheal, has not reached a post-menopausal state (≥12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).
  * Examples of contraceptive methods with a failure rate of ≤1% per year include bilateral tubal ligation, male sterilization, established proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.Hormonal contraception methods must be supplemented by a barrier method.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse), or use a condom, and agreement to refrain from donating sperm, as defined below:

  * With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 60 days after the last dose of mosunetuzumab and tocilizumab (if applicable) to avoid exposing the embryo. Men must refrain from donating sperm during this same period.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

* Inability to comply with all the study-related procedures, in the investigator's judgement.
* FL grade 3B or transformed FL
* Patients not meeting criteria for systemic therapy as outlined in section 6.1 and Appendix 4
* Patients unfit for chemoimmunotherapy for reasons including, but not limited to, advanced age and medical comorbidities
* FL presenting with isolated extra-nodal localizations, such as duodenal FL, cutaneous FL or FL of the testis
* Pediatric FL
* Prior anti-lymphoma therapy
* Prior solid organ transplantation
* Prior allogeneic stem cell transplantation within 5 years of FL diagnosis. Previously transplanted patients must be off all GVHD-related prophylaxis in order to be considered eligible.
* Current or prior central nervous system (CNS) lymphoma
* Current or past history of significant CNS disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease

  * Patients with a history of stroke who have not experienced a stroke or transient ischemic attack in the past 2 years and have no residual neurologic deficits as judged by the investigator are allowed
  * Patients with a history of epilepsy who have had no seizures in the past 2 years while not receiving any anti-epileptic medications are allowed
* Significant cardiovascular disease such as New York Heart Association Class III or IV cardiac disease [see Appendix 6], myocardial infarction within the last 6 months, unstable arrhythmias, or unstable angina
* Significant active pulmonary disease (e.g., bronchospasm or obstructive pulmonary disease)
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment, or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks prior to first mosunetuzumab administration
* Known or suspected chronic active Epstein-Barr Virus infection
* Serologic or PCR test results indicating acute or chronic HBV infection

  ° Patients whose HBV infection status cannot be determined by serologic test results (www.cdc.gov/hepatitis/hbv/pdfs/serologicchartv8.pdf) must be negative for HBV by PCR to be eligible for study participation.
* Acute or chronic HCV infection

  ° Patients who are positive for HCV antibody must be negative for HCV by PCR to be eligible for study participation.
* Serologic test results indicating HIV infection
* Administration of a live, attenuated vaccine within 4 weeks before first dose of study treatment or anticipation that such a live attenuated vaccine will be required during the study

  * Patients must not receive live, attenuated vaccines (e.g., FluMist®) while receiving study treatment or after the last dose until B-cell recovery to the normal ranges. Killed vaccines or toxoids should be given at least 4 weeks prior to the first dose of study treatment to allow development of sufficient immunity.
  * Inactivated influenza vaccination during influenza season and the COVID-19 vaccination at any time are allowed. Please see section 10.3.2 (permitted concomitant therapy) for additional guidance on SARS-CoV-2 vaccine administration and timing
  * Investigators should review the vaccination status of potential study patients being considered for this study and follow the U.S. Centers for Disease Control and Prevention guidelines for adult vaccination with any other non-live vaccines intended to prevent infectious diseases prior to study.
* Pregnant, lactating, or intending to become pregnant during the study or within 3 months after the last dose of mosunetuzumab and 3 months after the last dose of tocilizumab (if applicable)

  ° Women who are not postmenopausal (≥12 months of non-therapy-induced amenorrhea) or surgically sterile (removal of ovaries and/or uterus) must have a negative serum pregnancy test result within 14 days prior to initiation of study drug. If a serum pregnancy test has not been performed within 14 days prior to receiving first study treatment, a negative urine pregnancy test result (performed within 7 days prior to study treatment) must be available.
* Radiation therapy, unless utilized for the sole purpose of acutely controlling symptomatic disease during the screening period. In this case, at least 2 weeks should lapse between the last radiation dose and the first mosunetuzumab administration and the patient must still have measurable disease outside the field of radiation prior to initiation of the study drug
* Recent major surgery within 4 weeks prior to first mosunetuzumab administration, except protocol-mandated procedures (e.g., tumor biopsies and bone marrow biopsies)
* History of autoimmune disease, including, but not limited to myocarditis, pneumonitis, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis

  * Patients with a remote history of, or well-controlled autoimmune disease, may be eligible to enroll after discussion with and confirmation by the PI.
  * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
  * Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible for this study.
  * Patients with a history of disease-related immune thrombocytopenic purpura or autoimmune hemolytic anemia may be eligible for this study.
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:
  * Rash must cover <10% of body surface area
  * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
  * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months.
* History of known HLH or suspected HLH in the opinion of the investigator
* History of confirmed progressive multifocal leukoencephalopathy (PML)
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy (or recombinant antibody-related fusion proteins)
* History of other malignancy, except:

  * Curatively treated basal cell carcinoma, squamous cell carcinoma of the skin, in situ cervical carcinoma, in situ prostatic neoplasia.
  * A malignancy treated with curative intent and in remission for at least 2 years prior to the first mosunetuzumab administration
* Receipt of systemic immunosuppressive medications (including but not limited to cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) with the exception of corticosteroid treatment ≤10 mg/day prednisone or equivalent within 2 weeks prior to first dose of mosunetuzumab. The following is permitted:

  * The use of up to 12 mg/day dexamethasone for up to 3 days as antiemetic therapy
  * The use of up to 1mg/kg of prednisone or equivalent for ≤7 days to control B symptoms
  * The use of inhaled corticosteroids
  * The use of mineralocorticoids for management of orthostatic hypotension
  * The use of physiologic doses of corticosteroids for management of adrenal insufficiency
  * The use of premedication corticosteroids prior to undergoing contrast-enhanced imaging studies, in patients who are allergic to contrast agents
* History of illicit drug or alcohol abuse within 12 months prior to screening, in the investigator's judgment
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's or PI's judgment, precludes the patient's safe participation in and completion of the study, or which could affect compliance with the protocol or interpretation of results

Cohort 2 only:

* Requirement fors ongoing treatment with a strong CYP3A inhibitor or inducer (see section 15.2.3.2)
* History of severe bleeding disorder such as hemophilia A, hemophilia B, von Willebrand disease, or history of spontaneous bleeding requiring blood transfusion or other medical intervention.
* History of intracranial hemorrhage ≤ 180 days before the first dose of study treatment
* Inability to swallow capsules clinically significant or gastrointestinal dysfunction such as demonstrated malabsorption syndrome, resection of the stomach or small bowel, bariatric surgery, symptomatic inflammatory bowel disease, or bowel obstruction.
* Consumption of one or more of the following within 3 days prior to the first dose of zanubrutinib:

  * Grapefruit or grapefruit products
  * Seville oranges, including marmalade containing Seville oranges
  * Star fruit (carambola)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2022-05-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Complete Respons/CR | Up to 1 year
  The primary objective of the study is to determine the rate of Complete Response/CR to single-agent SC mosunetuzumab according to the 2014 Lugano response criteria in participants with newly diagnosed Follicular Lymphoma in need of systemic therapy.

SECONDARY OUTCOMES:
Overall Response Rate/ORR | Up to 3 years
  Assess the Overall Response Rate/ORR after treatment with single-agent SC mosunetuzumab mosunetuzumab

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Falchi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - Georgetown University (Data Collection Only), Washington D.C., District of Columbia
  - Memorial Sloan Kettering at Basking Ridge Limited Protocol Activities, Basking Ridge, New Jersey
  - Hackensack Meridian Health (Data collection only), Hackensack, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk- Commack (Limited protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited protocol activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited protocol activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org